CLINICAL TRIAL: NCT06399575
Title: Characterizing the Repeatability and Reproducibility of Cardiovascular Responses to Hypoxic Apneas
Brief Title: Characterizing Hypoxic Apnea Intra-individual Repeatability
Acronym: CHAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00138947
Record Dates: First submitted 2024-04-21; First posted 2024-05-06 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Hypoxia; Apnea
Keywords: Repeatability; Reproducibility; Heart Rate
MeSH Terms: conditions — Hypoxia; Apnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apnea Following Isocapnic Hypoxia (Experimental)
  Interventions: Other: Apnea Following Isocapnic Hypoxia

INTERVENTIONS:
Other: Apnea Following Isocapnic Hypoxia — Decreasing end-tidal partial pressure of oxygen to 50 mmHg for five minutes, targeting 80-85% peripheral oxygen saturation. The end-tidal partial pressure of carbon dioxide will remain +1 mmHg above baseline levels. After five minutes of hypoxia, participants will complete an apnea.

SUMMARY:
Apneas (breath-holds) are increasingly being tested in human subjects to understand how the human body operates. Apneas decrease heart rate and increase blood pressure. These findings are driving current research into the effects of oxygen concentrations on the heart rate and blood pressure responses to apneas and the effect of breath-hold training on these responses. The interest in apnea research is three-fold:

1. Apneas are a nervous system stressor that can help researchers better understand the fundamental operation of the human body;
2. Elite divers can use findings from research to better their training and performance; and
3. The scientific understanding of apneas may translate to a better understanding of sleep apnea.

Despite this interest, little is known about the repeatability (the consistency within a single day) and reproducibility (the consistency between days) in the heart rate and blood pressure responses to apneas. This uncertainty limits the scientific interpretations from previous results. This study aims to determine the repeatability and reproducibility of heart rate and blood pressure responses to apneas. The goals of the study are:

1. To provide greater certainty to previous results; and
2. Inform best practices for future studies.

The study requires 20 healthy volunteers (10 females) and will measure heart rate, blood pressure, breathing parameters (expired gas concentrations, breathing volume and rate), and oxygen saturation. During the protocol, participants will complete two maximal voluntary apneas and five test apneas. The test apneas will all be the same length based on the longer of the two maximal voluntary apneas. Before each apnea, participants will also breathe low oxygen concentrations (hypoxia). Hypoxia provides a bigger decrease in heart rate during apneas than room air which makes it easier to see changes in heart rate responses between apneas (i.e., bigger signal-to-noise ratio). Participants will complete two identical test sessions on back-to-back days. The differences in heart rate and blood pressure responses to the five apneas within each session will determine repeatability and the differences between sessions will determine reproducibility. The investigators hypothesize that repeatability will be good and that repeatability within a session will be better than reproducibility between sessions.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 18-70

Exclusion Criteria:

* Having known cardiovascular or nervous system disease
* Low or high blood pressure (< 90/60 or >139/85, respectively)
* Taking any prescribed medications (other than oral contraceptives) that may affect cardiovascular system function
* Females who may be pregnant (self-reported)
* Involved in other studies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Heart Rate | Continuous collection during both visits (2 hours on back-to-back days). Data will be extracted during free breathing (1 minute average before each apnea) and during apneas (beat-by-beat extraction from the 10 beats preceding resumption of breathing).
  Electrocardiogram (lead II)

SECONDARY OUTCOMES:
Blood Pressure | Continuous collection during both visits (2 hours on back-to-back days). Data will be extracted during free breathing (1 minute average before each apnea) and during apneas (beat-by-beat extraction from the 10 beats preceding resumption of breathing).
  Finger Photoplethysmography
Cardiac Arrhythmias | Continuous collection during both visits (2 hours on back-to-back days). Data will be extracted during apneas (beat-by-beat observation from the 10 beats preceding the resumption of breathing).
  Assessed using electrocardiogram (lead II) by a trained researcher and reviewed by a cardiologist. Arrhythmias observable in lead II will be reported as a binary (i.e., yes/no) for each individual for each apnea. Example arrhythmias are premature atrial contractions and sinus pauses, though many more exist.
Peripheral Oxygen Saturation | Continuous collection during both visits (2 hours on back-to-back days). Data will be extracted during free breathing (1 minute average before each apnea) and during apneas (10 beats preceding the resumption of breathing to 1 minute after apnea end).
  Pulse Oximetry
Rating of Perceived Exertion | Apnea (immediately following apnea)
  Participants Rate the Effort of their Apnea using the Modified Borg Scale with scores from 1 to 10 with 1 representing no effort and 10 representing a maximal effort.
Apnea Duration | Start to end of apnea: apnea start determined using cessation of flow through the pneumotachometer, apnea end determined using respiratory belt strain gauge. Estimated apnea durations are 15-30 seconds.
  Time, in seconds, from the end of the last breath preceding the apnea to the resumption of breathing.

OTHER OUTCOMES:
End-Tidal Oxygen | Continuous collection during both visits (2 hours on back-to-back days). Data will be extracted during free breathing (1 minute average before apnea).
  S-3A/I Oxygen Analyzer & Model N-22M Sensor, AEI Technologies
End-Tidal Carbon Dioxide | Continuous collection during both visits (2 hours on back-to-back days). Data will be extracted during free breathing (1 minute average before apnea).
  CD-3A Carbon Dioxide Analyzer & P-61B Sensor
Minute Ventilation | Continuous collection during both visits (2 hours on back-to-back days). Data will be extracted during free breathing (1 minute average before apnea).
  Pneumotachometer

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Busch SA, Davies H, van Diepen S, Simpson LL, Sobierajski F, Riske L, Stembridge M, Ainslie PN, Willie CK, Hoiland R, Moore JP, Steinback CD. Chemoreflex mediated arrhythmia during apnea at 5,050 m in low- but not high-altitude natives. J Appl Physiol (1985). 2018 Apr 1;124(4):930-937. doi: 10.1152/japplphysiol.00774.2017. Epub 2017 Dec 21. PMID 29357505
- [Background] Busch SA, van Diepen S, Steele AR, Meah VL, Simpson LL, Figueroa-Mujica RJ, Vizcardo-Galindo G, Villafuerte FC, Tymko MM, Ainslie PN, Moore JP, Stembridge M, Steinback CD. Global REACH: Assessment of Brady-Arrhythmias in Andeans and Lowlanders During Apnea at 4330 m. Front Physiol. 2020 Jan 22;10:1603. doi: 10.3389/fphys.2019.01603. eCollection 2019. PMID 32038287
- [Background] Stanforth PR, Gagnon J, Rice T, Bouchard C, Leon AS, Rao DC, Skinner JS, Wilmore JH. Reproducibility of resting blood pressure and heart rate measurements. The HERITAGE Family Study. Ann Epidemiol. 2000 Jul;10(5):271-7. doi: 10.1016/s1047-2797(00)00047-8. PMID 10942874
- [Background] Hopkins WG. Measures of reliability in sports medicine and science. Sports Med. 2000 Jul;30(1):1-15. doi: 10.2165/00007256-200030010-00001. PMID 10907753
- [Background] Weir JP. Quantifying test-retest reliability using the intraclass correlation coefficient and the SEM. J Strength Cond Res. 2005 Feb;19(1):231-40. doi: 10.1519/15184.1. PMID 15705040

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-26): https://cdn.clinicaltrials.gov/large-docs/75/NCT06399575/Prot_SAP_000.pdf
  • Informed Consent Form (2024-06-25): https://cdn.clinicaltrials.gov/large-docs/75/NCT06399575/ICF_001.pdf